CLINICAL TRIAL: NCT00809744
Title: Vitamin D AND Cardiovascular Disease
Brief Title: Vitamin D AND Glucose Handling Evaluated by Glucose Clamp
Acronym: D-clamp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian Council on Cardiovascular diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UIT-ENDO-2008-GURI-2
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Insulin Sensitivity; Intraocular Pressure
MeSH Terms: conditions — Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cholecalciferol — capsules, 20 000IU, twice a week, 6 months duration

SUMMARY:
In this study the investigators want to compare glucose handling (insulin secretion and insulin sensitivity) in 100 persons with low and 50 persons with normal-high levels of vitamin D, using a hyperglycemic clamp technique, were sugar is given intravenously for 3 hours in order to keep the blood sugar level at 10 mmol/L. Those with low vitamin D levels will be randomized to treatment with vitamin D3 (cholecalciferol) 40 000 IU/week or placebo for 6 months before a new clamp is performed.

The study hypothesis is that persons with low vitamin D levels have impaired glucose handling which might be improved by vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* generally: Subjects are recruited from the 6th Tromsø Study
* cases: serum 25-hydroxyvitamin D-levels below the 10 percentile; low levels confirmed with new serum analyses.
* controls: serum 25-hydroxyvitamin D levels 80-95 percentile, normal-high levels confirmed with new serum analyses.

Exclusion Criteria:

* diabetes
* myocardial infarction or apoplexia
* active cancer during last 5 years
* history of kidney stone
* pregnancy or premenopausal without safe anticonception
* primary hyperparathyroidism
* systolic blood pressure >175 or diastolic blood pressure >105

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
insulin secretion and sensitivity as assessed by an hyperglycemic clamp | 6 months
intraocular pressure | 6 months

SECONDARY OUTCOMES:
telomer length | 6 months
25-hydroxyvitamin D and 1,25-dihydroxyvitamin D-levels | 6 months
serum calcium, PTH, phosphate | 6 months
inflammatory markers and lipids | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — Medical Dpt, University Hospital of Northern Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Grimnes G, Figenschau Y, Almas B, Jorde R. Vitamin D, insulin secretion, sensitivity, and lipids: results from a case-control study and a randomized controlled trial using hyperglycemic clamp technique. Diabetes. 2011 Nov;60(11):2748-57. doi: 10.2337/db11-0650. Epub 2011 Sep 12. PMID 21911741